CLINICAL TRIAL: NCT05726747
Title: Health-related Quality of Life Outcomes and Changes in Sarcopenia in Patients With Refractory Ascites
Brief Title: QOL and Sarcopenia in Patients With Ascites
Status: Recruiting | Type: Observational
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Principal Investigator, Michael C Soulen, MD, Director Interventional Oncology, Abramson Cancer Center at Penn Medicine
Other Study IDs: UPCC 22222
Record Dates: First submitted 2023-02-02; First posted 2023-02-14 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Ascites Hepatic; Ascites, Malignant
Keywords: ascites; sarcopenia
MeSH Terms: conditions — Ascites; Sarcopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Quality of Life surveys — QoL and sarcopenia assessments
  Other Names: Abdominal CT

SUMMARY:
Clinical data regarding quality of life in patients with refractory ascites is limited and preceded the development of newer questionnaires that may be more robust. One primary objective of this study is to study changes in quality in life in a prospective fashion using newer general and ascites-specific quality of life survey instruments specific to benign and malignant etiologies.

Sarcopenia is a condition that is prevalent in cancer and cirrhosis. Current data is retrospective and associative, evaluating heterogeneous patient populations at different stages within the timeline of refractory ascites. The other primary objective of this study is to study sarcopenia in a prospective fashion and to understand its kinetics once a patient develops refractory ascites.

Prospectively-obtained measures of deterioration in patient-reported outcomes and in muscle mass will form the basis for the next stage of investigation of interventions to mitigate these declines.

DETAILED DESCRIPTION:
Patients with refractory ascites defined as requiring >1 paracentesis within a 6 week period will be prospectively enrolled. The Patient-Reported Outcomes Measurement Information System (PROMIS-10) and ascites-specific (Ascites Q and Edmonton Symptom Assessment System: Ascites Modification) quality of life questionnaires will be obtained at baseline, then at 1-, 2-, 4- and 6 months. Sarcopenia will be assessed by muscle area measurement from a single CT image at the L4 level at baseline, 2- and 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Age >/=18
2. Eastern Cooperative Oncology Group (ECOG) performance score < 3
3. Refractory ascites due to cirrhosis or malignancy, requiring more than 1 therapeutic paracentesis in a 6 week period within 3 months of enrollment.
4. Capable of giving informed consent

Exclusion Criteria:

1. Life expectancy less than 3 months
2. Unable to participate in neuropsychological tests/questionnaires
3. Pregnant or nursing women. .

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 35-40 unique patients are seen by interventional radiology in the Perelman Center for Advanced Medicine or the Hospital of the University of Pennsylvania for a therapeutic paracentesis per month in an outpatient setting. Approximately half of these patients (~20 per month) meet criteria for refractory ascites requiring frequent large volume paracentesis (i.e. more than 1 therapeutic paracentesis in a 6 week period).
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2023-05-23 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Health-Related Quality of Life scores as measured by the PROMIS-10 questionnaire | 6 months
  Patient-Reported Outcomes Measurement Information System (PROMIS-10) survey scores physical and mental health on a 4-20 point scale which are combined into an overall score with higher scores reflecting better quality of life.
Sarcopenia as measured by psoas, paraspinal, and total abdominal wall muscle areas | 6 months
  assessed by a limited CT scan of the abdomen at the level of L4. Cross-sectional muscle area is measured.

SECONDARY OUTCOMES:
Ascites-specific QOL scores as measured by the Ascites Q for patients with cirrhotic ascites. | 6 months
  Ascites Q asks 11 questions on a 2-11 scale. Total is normalized to a 0-100 point scale with higher score reflecting worse symptoms.
Ascites-specific QOL scores as measured by the Edmonton Symptom Assessment System: Ascites Modification for patients with malignant ascites, | 6 months
  11 questions on a 0-10 scale, total score range 0-110 with higher score reflecting worse symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Soulen, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania Perelman School of Medicine, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No